CLINICAL TRIAL: NCT05172583
Title: Nursing Intervention to Reduce Incidence and Duration of Delirium in Patients in Intensive Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Surcolombiana (Other)
Collaborators: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 53487
Record Dates: First submitted 2021-09-30; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-09

CONDITIONS: Delirium
Keywords: Delirium; Intensive Care Units; Disease Prevention; Evaluation of the Efficacy-Effectiveness of Interventions; Non-pharmacological interventions
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Intervention Model Description: Participants will be recruit upon admission to the ICU, patients and family members are asked to sign the informed consent and confidentiality agreement. The Assignment to the groups will be random. All interventions will be performed and will be adjusted according to the patient's condition. If the patient is recruited while under the effects of sedation, they will be asked to sign the informed consent when she is conscious; if she does not wish to participate, the withdrawal will be completed, and she will be excluded from the study. Follow-up will be done each shift, where the outcome variables will be measured and recorded in an established format.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be triple-blind, since the participants and their relatives, the research assistant who measures the outcome variables, and who performs the information analysis process, will not know the assignment of the study, control and intervention groups, due to They will be named by categories coded by the research assistant who performs the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The control groups will receive the nursing interventions that are performed daily in the adult ICU
  Interventions: Behavioral: Control
- Experimental (Experimental): Interventions for this group are based on the Dynamic Symptom Model and scientific evidence
  Interventions: Behavioral: Interventions to reduce delirium based on DSM and scientific evidence

INTERVENTIONS:
Behavioral: Control — The control groups will receive the nursing interventions that are performed daily in the adult ICU. These are orientation in time, space, and place, accompaniment of the family for two hours in the morning and two hours in the afternoon, physical therapy once a day according to the patient's condition, medication with conscious sedation, and progressive reduction analgesics. opioids and benzodiazepines.
  Arms: Control
Behavioral: Interventions to reduce delirium based on DSM and scientific evidence — The interventions are designed from the structure of the Dynamic Symptoms Model (DSM), taking into account the antecedents of delirium, physiological such as the medical condition of mechanical ventilation and pain, and drug treatment with sedatives and analgesics; the psychological, social, and spiritual antecedents with stimulation in the values, life experience, personality and spirituality, and the environmental antecedents with an adaptation of the physical conditions of the ICU. In addition, previous experience with identification and care of concomitant symptoms such as fear, confusion, restlessness, loneliness, and discomfort, and with the measurement and classification of the trajectory of delirium when it occurs, will also be considered. The interventions follow the scientific evidence, mainly from the ABCDEF bundle. All interventions are non-pharmacological.
  Arms: Experimental

SUMMARY:
Introduction: Delirium is a cognitive alteration of acute onset and fluctuating course, characterized by the reduced capacity to pay attention to the environment, memory impairment, disorientation, language, and perception alteration. Its incidence varies between 20 and 90% in ICU patients. It shows high variability in both incidence and typology, representing a phenomenon of great interest to nursing, who can make timely interventions.

General objective: To determine the effectiveness of nursing interventions based on the Dynamic Symptoms Model and scientific evidence, compared to daily care, for reducing the incidence and duration of delirium in people hospitalized in the adult ICU.

Methodology: Study with a quantitative approach, experimental design of the type Randomized Controlled Clinical Trial of parallel groups, phase III in which the effectiveness and safety of the intervention designed in a particular population are evaluated, such as the ICU population, who are older risk of developing delirium. The sample will be 71 people for the intervention group and 142 for the control group, with a 2: 1 ratio.

Expected outcome: The primary results are: reduce the incidence and duration of delirium in ICU patients, and the secondary outcomes are: shorter ICU stay, mechanical ventilation, use of physical restraints, less pain intensity, and more days in RASS between -2 and + 1.

Risk: Greater than the minimum.

DETAILED DESCRIPTION:
Framework Delirium epidemiology

Delirium is a cognitive alteration, with an acute onset and fluctuating course, characterized by a reduced ability to pay attention to the environment, memory impairment, disorientation, language and perception disturbances(1). Its occurrence varies between 20 and 90% in people hospitalized in the Intensive Care Unit (ICU) (2,3), with a duration between 1 and 5 days (2,3). Its hypoactive typology is frequent between 5 and 71.5% of the cases, hyperactive between 5.1 and 14%, and mixed between 5.1 and 89%. Its shows high variability in both incidence and typology, representing a phenomenon of great interest to nursing, who can make timely interventions.

Various studies have found that the etiology of delirium is associated with predisposing and precipitating factors. Among the predisposing factors, there is age between 50 and 70 years (4). Also chronic kidney disease, cerebrovascular disorders and a previous history of delirium, cognitive dysfunction, depression, dementia, dependence on psychoactive substances and / or alcohol, postoperative states, arterial hypertension, disease severity, elevated blood urea nitrogen and creatinine, sodium and hyperthermia(4).

Among the precipitating factors of delirium are mechanical ventilation (5), benzodiazepines (2), low scores in the RASS scale (5), pain, stress, interruption of the sleep-wake cycle, physical immobilizations, and medical devices such as urinary catheter and central venous catheter. These factors are specific to the environment and ICU treatment and increase the risk of delirium, regardless of the presence or absence of predisposing factors. However, the precipitating factors are modifiable according to the diagnosis and evolution of the patient.

Its impact is highly negative since it increases the days of mechanical ventilation, of consciousness in deep sedation (5), stay and mortality in ICU and hospital (2), of the use of physical restraints accelerates the transition to dementia and reduces cognitive recovery, and physical functionality(3). For this reason, the American Guidelines of 2013 and 2018 and German of 2015 for the management of agitation, pain, and delirium, recommend monitoring and preventing it through mainly non-pharmacological measures, which is part of the strategy of humanization of care in the ICU.

The high incidence and consequences of delirium in people hospitalized in the ICU continues to be worrying; however, the detection of precipitating factors suggests alternative measures that make the environment and care modifiable, to reduce the incidence and duration of delirium. On the other hand, the predisposing factors of delirium suggest a baseline or possible confounding variables to detect and control in the present study.

Nursing has a dominant role in the approach to delirium. The assessment and Nurses' interventions are essential to prevent and treat delirium. Nurses are leaders in clinical decision-making; since they constantly evaluate people's conditions and their clinical results, they are the ones who have the most and timely communication with patients. von Rueden et al. (5) add that. Therefore, nursing interventions can reduce the risk of delirium, the length of stay in ICU, mortality, and long-term impairment of cognition.

Main propositions:

* Initial measures to address delirium include the identification and correction of precipitating cause. In addition, non-pharmacological interventions can prevent delirium.
* A variety of ICU care processes influence delirium, most of which are modifiable.
* Through the development and implementation of evidence-based interventions, it is possible to reduce the incidence and duration of delirium.

Main Gaps:

The incidence of delirium in the ICU remains high (20-90%) and its harmful consequences, although evidence-based packages prevent it.

- Health professionals, including nurses, have naturalized delirium in ICU patients, which has reduced the possibilities of prevention.

Justification

The onset of delirium in people in the ICU remains high in European, Asian, and American countries; it ranges between 20 and 90% (2). In Colombia, it ranges between 20.2 and 28% (6). It is associated with predisposing and precipitating factors. The latter is related to the care provided in the ICU, which is mostly modifiable. Its consequences are loss of factual memory, increased ICU and hospital stay, medical care costs, days of mechanical ventilation, and even mortality (2). Not only patients are affected, but also their families and the health system in general. Therefore, it is pertinent to develop strategies that mitigate their incidence and impact.

Although effective interventions are found in the scientific evidence to prevent and treat delirium, its incidence remains high, which justifies the need to develop and implement non-pharmacological interventions early. In this regard, in this study, in addition to implementing interventions based on scientific evidence, they will be designed from a theoretical perspective, such as the Dynamic Symptoms Model, which offers support to the approach method, since it provides a structure congruent with the phenomenon, in turn, giving, the novelty in the development of interventions, because it includes elements not addressed in other studies such as psychological, spiritual, social, environmental antecedents, previous and concomitant experiences and symptoms, as well as the broad participation of the family in all interventions.

It is feasible to carry out this research because there is access to the population and institution of study, with thematic and methodological advice and the academic and ethical support of the National University of Colombia. Furthermore, it is feasible because it is a phenomenon susceptible to measurement and intervention, there are validated tools, and the interventions will solve a problem in nursing practice.

Research question: What is the effectiveness of nursing interventions based on the Dynamic Symptom Model and scientific evidence, compared to daily care, to reduce the incidence and duration of delirium in people hospitalized in the adult ICU?

General objective: To determine the effectiveness of nursing interventions based on the Dynamic Symptom Model and scientific evidence, compared to daily care, for reducing the incidence and duration of delirium, in people hospitalized in the adult ICU.

Specific objectives according to study phases:

Phases I. Design of the intervention

* Design the nursing intervention based on the conceptual structure of the Dynamic Symptoms Model and scientific evidence to reduce the incidence and duration of delirium in patients in intensive care.
* Analyze the feasibility, viability, and barriers of the designed intervention through validation by experts working in the institution.

Phase II. Evaluation of the intervention

* Characterize demographically and clinically the people participating in the study.
* Compare the intervention designed, versus daily care, in reducing the incidence and duration of delirium and other clinical outcomes (reduction in days of mechanical ventilation and stay in the ICU, the presence and intensity of pain, the use of physical restrictions, and the improvement of the state of consciousness).

Hypothesis

Study hypothesis: The nursing intervention based on the Dynamic Symptoms Model and scientific evidence reduce incidence and duration of delirium in people hospitalized in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* People admitted to the adult intensive care unit
* People over 18 years of age.
* People who are agree to participate in the study by signing the informed consent.
* People who have no delirium at the time of recruitment (CAM - negative ICU).

Exclusion Criteria:

* People with any cognitive disorder or neurosurgical pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive state, presence or absence of delirium with Confusion Assessment Method for the Intensive Care Unit CAM-ICU scale | Through ICU length of stay, an average of 8 days.
  The possible results are positive or negative for delirium

SECONDARY OUTCOMES:
Fluctuations in consciousness with Richmond Agitation-Sedation Scale (RASS). | Through ICU length of stay, an average of 8 days.
  The Richmond Agitation-Sedation Scale measures the sedation and agitation level in patient in Intensive care unit. Its possible results are: -5 unarousable, -4 deep sedation, -3 moderate sedation, -2 light sedation, -1 drowsy, 0 alert and calm, +1 restless, +2 agitated, +3 very agitated, and +4 combative.
Changes in the Pain intensity. with Campbell scale in non-communicative critical patients, and Visual Analog Scale (VAS) in communicative critical patients. | Through ICU length of stay, an average of 8 days.
  Campbell scale measures the pain intensity. Its results are: 0 without pain, 1-3 between mild and moderated pain, 4-6 between moderate and severe pain, and >6 intensive pain. The possible results of Visual Analog Scale are 0 no pain, 1-3 mild pain, 4-6 between moderate and severe pain, 7-9 very severe pain, 10 worst pain possible.
  Campbell scale measures the pain intensity. Its results are: 0 without pain, 1-3 between mild and moderated pain, 4-6 between moderate and severe pain, and >6 intensive pain. The possible results of Visual Analog Scale are 0 no pain, 1-3 mild pain, 4-6 between moderate and severe pain, 7-9 very severe pain, 10 worst pain possible.
length of stay in ICU | Through ICU length of stay, an average of 8 days.
  length of stay in ICU
Mechanical ventilation | Through ICU length of stay, an average of 8 days
  Number of Mechanical ventilation days
Physical restrictions | Through ICU length of stay, an average of 8 days.
  Number with physical restrictions days

CONTACTS AND LOCATIONS:
Overall Officials: Ángela M Henao Castaño, PhD, Study Director — Universidad Nacional de Colombia; Dolly O Arias Torres, PhD, Study Chair — Universidad Surcolombiana
Locations (1):
- Hospital Universitario Hernando Moncaleano Perdomo, Neiva, Huila Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vahia VN. Diagnostic and statistical manual of mental disorders 5: A quick glance. Indian J Psychiatry. 2013 Jul;55(3):220-3. doi: 10.4103/0019-5545.117131. No abstract available. PMID 24082241
- [Result] Mitchell ML, Kean S, Rattray JE, Hull AM, Davis C, Murfield JE, Aitken LM. A family intervention to reduce delirium in hospitalised ICU patients: A feasibility randomised controlled trial. Intensive Crit Care Nurs. 2017 Jun;40:77-84. doi: 10.1016/j.iccn.2017.01.001. Epub 2017 Feb 27. PMID 28254205
- [Result] Lee A, Mu JL, Chiu CH, Gin T, Underwood MJ, Joynt GM. Effect of motor subtypes of delirium in the intensive care unit on fast-track failure after cardiac surgery. J Thorac Cardiovasc Surg. 2018 Jan;155(1):268-275.e1. doi: 10.1016/j.jtcvs.2017.08.139. Epub 2017 Sep 30. PMID 29110954
- [Result] Park SA, Tomimaru Y, Shibata A, Miyagawa S, Noguchi K, Dono K. Incidence and Risk Factors for Postoperative Delirium in Patients After Hepatectomy. World J Surg. 2017 Nov;41(11):2847-2853. doi: 10.1007/s00268-017-4079-3. PMID 28608014
- [Result] Von Rueden KT, Wallizer B, Thurman P, McQuillan K, Andrews T, Merenda J, Son H. Delirium in Trauma Patients: Prevalence and Predictors. Crit Care Nurse. 2017 Feb;37(1):40-48. doi: 10.4037/ccn2017373. PMID 28148613
- [Result] Girard TD, Pandharipande PP, Ely EW. Delirium in the intensive care unit. Crit Care. 2008;12 Suppl 3(Suppl 3):S3. doi: 10.1186/cc6149. Epub 2008 May 14. PMID 18495054
- [Result] Ely EW. The ABCDEF Bundle: Science and Philosophy of How ICU Liberation Serves Patients and Families. Crit Care Med. 2017 Feb;45(2):321-330. doi: 10.1097/CCM.0000000000002175. PMID 28098628